CLINICAL TRIAL: NCT01291225
Title: Safe Play Areas for Ross County Kids Project
Acronym: SPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Gary A. Smith, PI, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB10-00368
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Other Specified Personal Exposures and History Presenting Hazards to Health; Knowledge, Attitudes, Practice; Fall Involving Playground Equipment, Occurrence on Farm
Keywords: playgrounds; farms; injury prevention; safety knowledge, attitudes and practices; safe play; rural
MeSH Terms: conditions — Behavior | interventions — Growth and Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Playground (Other): The playground arm of the study will consist of playground audits and KAP surveys about playground safety in both Chillicothe and Circleville, Ohio.
  The intervention is Playground Safety Renovations and Development.
  Interventions: Other: Playground renovation and development; Behavioral: Educational campaign
- Farms (Other): The Farm Arm will consist of farm audits with safety checklists and KAP surveys about farm safety. The intervention is a Safety Educational Campaign.
  Interventions: Behavioral: Educational campaign

INTERVENTIONS:
Other: Playground renovation and development — Playgrounds in Chillicothe will be renovated based on priorities determined by audits.
  Arms: Playground
Behavioral: Educational campaign — Educational materials will be developed and distributed in Ross County.

SUMMARY:
Specific Aim 1 - In collaboration with partners in Ross County, renovate and develop playgrounds in Chillicothe.

Specific Aim 2 - In collaboration with partners in Ross County, promote safe play and play areas for children on farms.

DETAILED DESCRIPTION:
Injury is the leading cause of mortality and morbidity among children in the United States. Because children spend much of their time playing, it is important that they have safe play environments where they can challenge themselves and develop physically, mentally, and socially. The SPARK Project will focus its intervention in Ross County, Ohio, an area with more than 930 farms. Prior to this project, relatively little has been done to promote the prevention of injuries to children who live and play on farms.

The specific aims of this project are as follows:

* In collaboration with partners in Ross County, renovate and develop playgrounds in Chillicothe, Ohio.
* In collaboration with partners in Ross County, promote safe play areas for children on farms.

The SPARK Project will employ a multi-faceted approach to injury prevention, centered on community partnership and collaboration. Utilizing methodology that was successfully developed and implemented as part of the Community Action for Playground Safety (CAPS) Program in Columbus, the SPARK Project will combine both active and passive injury prevention strategies to reduce playground and play-related farm injuries to children in Ross County.

ELIGIBILITY:
Inclusion Criteria:

* For playgrounds

  * must be seen at Adena Medical Center or Pickaway Pediatrics
  * must be the parent of a child younger than 6 years of age
  * must live in Chillicothe (if recruited at Adena) or Circleville (if recruited at Pickaway Peds)
  * must be English speaking
  * must be at least 18 years old
* For farms

  * must self-identify as living on a farm
  * must have a child younger than 6 years of age
  * must live in Ross county or Pickaway county
  * must be English speaking
  * must be at least 18 years old

Exclusion Criteria:

* Participants can only enroll in one study at a time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Smith, MD, DrPH, Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- The Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Playground: The playground arm of the study will consist of playground audits and KAP surveys about playground safety in both Chillicothe and Circleville, Ohio.
- Farms: The Farm Arm will consist of farm audits with safety checklists and KAP surveys about farm safety.
Period: Overall Study
Arm/Group | Playground | Farms
Started | 151 | 160
Completed | 66 | 121
Not Completed | 85 | 39
Not completed — Lost to Follow-up | 85 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Playground | Farms | Total
Number analyzed (Participants) | 151 | 160 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 151 | 160 | 311
  >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 151 | 160 | 311
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 129 | 262
  Male | 18 | 31 | 49
Region of Enrollment [Number; unit: participants]
  United States | 151 | 160 | 311

OUTCOME MEASURES:

1. Primary Outcome: Change in Playground Hazards
Description: The investigators hypothesize that the decrease in the number of identified playground hazards (comparing each playground to itself from the year 1 baseline survey to the year 3 follow-up survey utilizing a playground hazards checklist) will be significantly greater for the intervention playgrounds compared with non-intervention playgrounds in Circleville, Pickaway Co. The percentage increase in the number of playgrounds with adequate safety surfacing will be used as a proxy for playground hazardousness.
Time Frame: Year 1 baseline to year 3 follow-up
Measure: Number; unit: % increase playgrounds w/surfacing
Arm/Group | Playground | Farms
Number analyzed (Participants) | 66 | 121
% increase playgrounds w/surfacing
  Intervention | 50 | 0
  Control | 0 | 0

2. Secondary Outcome: Playground and Farm Safety Knowledge, Attitudes and Practices Composite Scores
Description: The investigators hypothesize that the improvement in the playground safety Knowledge, Attitudes, and Practices (KAP) survey composite scores and farm audits from the baseline in year 1 to the follow-up in year 3 will be significantly greater for parents residing in Ross County than for parents in the non-intervention counties (Morrow and Pickaway).The playground safety KAP survey consisted of 7 items and individuals could receive a summed score of 0-7, with a score of 7 indicating mastery of the material.
Time Frame: Year 1 baseline to Year 3 follow-up
Measure: Mean (Standard Deviation); unit: composite score
Groups:
- Playground--Chillicothe; Playground--Circleville: The playground arm of the study will consist of playground audits and KAP surveys about playground safety in both Chillicothe and Circleville, Ohio.
- Farms--Ross County; Farms--Pickaway/Morrow Counties: The Farm Arm will consist of farm audits with safety checklists and KAP surveys about farm safety.
Arm/Group | Playground--Chillicothe | Playground--Circleville | Farms--Ross County | Farms--Pickaway/Morrow Counties
Number analyzed (Participants) | 25 | 41 | 55 | 66
composite score | 5.2 (0.7638) | 5.1 (0.6149) | NA (NA) — Farm audtis were not completed | NA (NA) — Farm audits were not completed

ADVERSE EVENTS:
Arm/Group | Playground | Farms
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/160
Other Adverse Events (participants affected / at risk) | 0/151 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes